CLINICAL TRIAL: NCT06119113
Title: Evaluation of Wound Site Infection,Early and Late Wound Healing and Cosmetic Results of Vicryl ,Monocryl and Prolene Suture Materials Used in Pfannenstiel Skin Incision in Caesarean Section
Brief Title: Evaluation of Wound Infection Rates and Cosmetic Results of Different Suture Materials in Cesarean Skin Incision
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ayşenur Çalış Özbayram (Other Government)
Responsible Party: Sponsor-Investigator, Ayşenur Çalış Özbayram, Gynecology And Obstetrics Doctor, Başakşehir Çam & Sakura City Hospital
Organization: Başakşehir Çam & Sakura City Hospital (Other Government)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: basaksehircamvesakurasehirh
Record Dates: First submitted 2023-09-27; First posted 2023-11-07 (Actual); Results first posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Cesarean Section; Infection; Scar
Keywords: suture material; Caesarean section skin scar; Pfannenstiel
MeSH Terms: conditions — Infections; Cicatrix

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 (Vicryl suture™(Polyglactin 910)) (Active Comparator): The group whose skin incision was closed with Vicryl suture™ (Polyglactin 910) from patients who had cesarean section for the first time
  Interventions: Other: Evaluation of the wound infection at the 10th day post-op check-up among all groups; Other: Evaluation of the cosmetic results of the incision line at the 2nd month post-op check-up among all groups; Other: Evaluation of the cosmetic results of the incision line at the 6th month post-op check-up among all groups
- Group 2 (Prolene suture™(polypropylene)) (Active Comparator): The group whose skin incision was closed with Prolene suture™ (polypropylene) from patients who had cesarean section for the first time
  Interventions: Other: Evaluation of the wound infection at the 10th day post-op check-up among all groups; Other: Evaluation of the cosmetic results of the incision line at the 2nd month post-op check-up among all groups; Other: Evaluation of the cosmetic results of the incision line at the 6th month post-op check-up among all groups
- Group 3 (Monocryl suture™ (Polyglecaprone 25)) (Active Comparator): The group whose skin incision was closed with Tekmon suture™ (Polyglecaprone 25) from patients who had cesarean section for the first time
  Interventions: Other: Evaluation of the wound infection at the 10th day post-op check-up among all groups; Other: Evaluation of the cosmetic results of the incision line at the 2nd month post-op check-up among all groups; Other: Evaluation of the cosmetic results of the incision line at the 6th month post-op check-up among all groups

INTERVENTIONS:
Other: Evaluation of the wound infection at the 10th day post-op check-up among all groups — Discharge, redness, increased temperature, and dehiscence were accepted as wound infection.
  Other Names: Post-op Control
Other: Evaluation of the cosmetic results of the incision line at the 2nd month post-op check-up among all groups — The cosmetic outcome of wound site scar healing was evaluated with two different scales. The Patient and Observer Assessment Scale (POSAS) is a questionnaire developed to assess scar quality. The investigator scores six items: vascularization, pigmentation, thickness, surface roughness, elasticity, and surface area. The participant scores six items: pain, itching, color, thickness, relief, and flexibility. All items are scored on a 10-point multiple scale; A score of 1 is given when the scar characteristic is similar to 'normal skin' and a score of 10 is given when it reflects the 'worst scar'. All items are summed to determine the total scar score; a higher score represents worse scar quality. The Vancouver scar scale (VSS) consists of four variables: vascularity, height (thickness), elasticity and pigmentation. The total score ranges from 0 to 14, with a score of 0 reflecting normal skin.
  Other Names: Post-op Control
Other: Evaluation of the cosmetic results of the incision line at the 6th month post-op check-up among all groups — The cosmetic outcome of wound site scar healing was evaluated with two different scales. The Patient and Observer Assessment Scale (POSAS) is a questionnaire developed to assess scar quality. The investigator scores six items: vascularization, pigmentation, thickness, surface roughness, elasticity, and surface area. The participant scores six items: pain, itching, color, thickness, relief, and flexibility. All items are scored on a 10-point multiple scale; A score of 1 is given when the scar characteristic is similar to 'normal skin' and a score of 10 is given when it reflects the 'worst scar'. All items are summed to determine the total scar score; a higher score represents worse scar quality. The Vancouver scar scale (VSS) consists of four variables: vascularity, height (thickness), elasticity and pigmentation. The total score ranges from 0 to 14, with a score of 0 reflecting normal skin.
  Other Names: Post-op Control

SUMMARY:
Our primary aim is to determine the most beneficial suture in order to reduce complications due to skin incision in common surgeries such as cesarean section, and our secondary aim is to evaluate the suture material used in terms of cosmetic results and participant preference.

DETAILED DESCRIPTION:
Patients who met the inclusion criteria among patients who had a cesarean delivery (January 2023-June 2023) in our hospital within a 6-month period will be included in the study. Patients included in the study will be randomized and divided into three randomized groups as Vicryl (Polyglactin 910), Monocryl (Polyglecaprone 25) and Prolene (polypropylene) to be administered. Each cesarean section technique will be left to the discretion of the surgeon performing the operation, and cefazolin 2 g will be administered prophylactically half an hour before each procedure in our clinic. In all cases, a Pfannenstiel skin incision will be made 2 cm above the pubic symphysis. Following delivery of the fetus, the uterus, peritoneum, and fascia will be closed in sequence. The skin will be sealed with Vicryl (Polyglactin 910), Monocryl (Polyglecaprone 25), and Prolene (polypropylene) according to randomization. The dressing will be removed on the first day after the operation and the patients will be discharged on the second post-op day if there is no problem after the operation. Patients will be called for control on the 10th , 60th and 120th days of pos op. If the post op 10th day is deemed appropriate, the sutures of the patients in the prolene suture group will be removed. All groups that come to the control will be evaluated with the patient and the observer doctor by the patient and observer rating scale (POSAS) and the Vancouver Scar Scale (VSS).

The Patient and Observer Rating Scale (POSAS) is a questionnaire developed to assess scar quality. It consists of a five-observer and six-patient scale (Observer and Patient Scales) according to the rating scale based on clinically relevant scar characteristics [ Draaijers LJ, 2004 , Van de Kar AL, 2005]. Observer ; scores six items: vascularization, pigmentation, thickness, surface roughness, flexibility, and surface area. Patient ; it scores six items: pain, itching, color, thickness, relief and flexibility [Van de Kar AL , 2005]. All included items are scored on a multiple 10-point scale where 1 point is given when the wound feature is similar to 'normal skin' and 10 points are awarded when it reflects the 'worst scar'. All items are summed to determine the total scar score, with a higher score representing worse scar quality.

The Vancouver scar scale (VSS) consists of four variables: vascularity, height (thickness), elasticity, and pigmentation. The total score ranges from 0 to 14, with a score of 0 reflecting normal skin

ELIGIBILITY:
Inclusion Criteria:

* 18-45 years old
* Patients who had a primary cesarean section at our >37w hospital
* Patients with a Pfannenstiel incision closed subcutaneously

Exclusion Criteria:

* Women <18 years and >45 years old
* Those with a history of keloid
* Suprapubic incision due to previous surgery
* Signs of infection at or near the incision during cesarean section
* Known hypersensitivity to any of the suture materials used
* Having a medical condition that causes immunosuppression, such as DM, chronic corticosteroid use
* Failure to obtain informed consent from the patient

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 300 (Actual)
Dates: Start 2023-02-22 (Actual); Primary Completion 2023-07-22 (Actual); Study Completion 2023-10-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ayşenur ÇALIŞ ÖZBAYRAM, Principal Investigator — yok
Locations (1):
- Başakşehir Çam Ve Sakura Şehir Hastanesi, Istanbul, Başakşehir, Turkey (Türkiye)

REFERENCES:
- [Background] Koroglu N, Temel Yuksel I, Aslan Cetin B, Aytufan Z, Deniz N, Akca A, Yetkin Yildirim G, Yuksel A. Skin closure at cesarean section, polypropylene versus polyglactin 910: a randomized controlled study. J Matern Fetal Neonatal Med. 2022 Mar;35(6):1088-1092. doi: 10.1080/14767058.2020.1743654. Epub 2020 Mar 30. PMID 32228099
- [Background] Cromi A, Ghezzi F, Gottardi A, Cherubino M, Uccella S, Valdatta L. Cosmetic outcomes of various skin closure methods following cesarean delivery: a randomized trial. Am J Obstet Gynecol. 2010 Jul;203(1):36.e1-8. doi: 10.1016/j.ajog.2010.02.001. Epub 2010 Apr 24. PMID 20417924
- [Result] Buresch AM, Van Arsdale A, Ferzli M, Sahasrabudhe N, Sun M, Bernstein J, Bernstein PS, Ngai IM, Garry DJ. Comparison of Subcuticular Suture Type for Skin Closure After Cesarean Delivery: A Randomized Controlled Trial. Obstet Gynecol. 2017 Sep;130(3):521-526. doi: 10.1097/AOG.0000000000002200. PMID 28796687
- [Result] Byrne M, Aly A. The Surgical Suture. Aesthet Surg J. 2019 Mar 14;39(Suppl_2):S67-S72. doi: 10.1093/asj/sjz036. PMID 30869751

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Inclusion Criteria:
  * 18-45 years old
  * Patients who had a primary cesarean section at 37w
  * Patients with a Pfannenstiel incision closed subcutaneously
Groups:
- Group 1 (Vicryl Suture™(Polyglactin 910)): The group whose skin incision is closed with Vicryl suture™ (Polyglactin 910) Evaluation of wound infection at the 10th postoperative day control: Discharge, redness, temperature increase and opening were accepted as wound infection.Evaluation of the cosmetic results of the incision line in all groups at the 2nd and 6th month postoperative controls: The cosmetic results of wound healing are two different It was evaluated with a scale. The Patient and Observer Assessment Scale (POSAS) is a questionnaire developed to evaluate scar quality. The researcher scores six items: vascularization, pigmentation, thickness, surface roughness, elasticity, and surface area. The participant scores six items: pain, itching, color, thickness, relief, and flexibility. All items are scored on a 10-point multiple scale; 1 point is given when the scar characteristic resembles 'normal skin', and 10 points are given when it reflects the 'worst scar'. All items are summed to determine the total scar score; a higher score represents worse scar quality. The Vancouver scar scale (VSS) consists of four variables: vascularity, height (thickness), elasticity and pigmentation. The total score ranges from 0 to 14, with a score of 0 reflecting normal skin.
- Group 2 (Prolene Suture™(Polypropylene)): The group whose skin incision is closed with Prolene suture™ (polypropylene) Evaluation of wound infection at the 10th postoperative day control: Discharge, redness, temperature increase and opening were accepted as wound infection. Evaluation of the cosmetic results of the incision line in all groups at the 2nd and 6th month postoperative controls: The cosmetic results of wound healing are two different It was evaluated with a scale. The Patient and Observer Assessment Scale (POSAS) is a questionnaire developed to evaluate scar quality. The researcher scores six items: vascularization, pigmentation, thickness, surface roughness, elasticity, and surface area. The participant scores six items: pain, itching, color, thickness, relief, and flexibility. All items are scored on a 10-point multiple scale; 1 point is given when the scar characteristic resembles 'normal skin', and 10 points are given when it reflects the 'worst scar'. All items are summed to determine the total scar score; a higher score represents worse scar quality. The Vancouver scar scale (VSS) consists of four variables: vascularity, height (thickness), elasticity and pigmentation. The total score ranges from 0 to 14, with a score of 0 reflecting normal skin.
- Group 3 (Monocryl Suture™ (Polyglecaprone 25)): The group whose skin incision is closed with Tekmon suture™ (Polyglecaprone 25) Evaluation of wound infection at the 10th postoperative day control: Discharge, redness, temperature increase and opening were accepted as wound infection. Evaluation of the cosmetic results of the incision line in all groups at the 2nd and 6th month postoperative controls: The cosmetic results of wound healing are two different It was evaluated with a scale. The Patient and Observer Assessment Scale (POSAS) is a questionnaire developed to evaluate scar quality. The researcher scores six items: vascularization, pigmentation, thickness, surface roughness, elasticity, and surface area. The participant scores six items: pain, itching, color, thickness, relief, and flexibility. All items are scored on a 10-point multiple scale; 1 point is given when the scar characteristic resembles 'normal skin', and 10 points are given when it reflects the 'worst scar'. All items are summed to determine the total scar score; a higher score represents worse scar quality. The Vancouver scar scale (VSS) consists of four variables: vascularity, height (thickness), elasticity and pigmentation. The total score ranges from 0 to 14, with a score of 0 reflecting normal skin.
Period: Overall Study
Arm/Group | Group 1 (Vicryl Suture™(Polyglactin 910)) | Group 2 (Prolene Suture™(Polypropylene)) | Group 3 (Monocryl Suture™ (Polyglecaprone 25))
Started | 100 | 100 | 100
Post op 10th Day Check-up | 92 | 95 | 96
Post op 2nd Month Check-up | 85 | 87 | 79
Post op 6st Month Check-up | 85 | 87 | 79
Completed | 85 | 87 | 79
Not Completed | 15 | 13 | 21
Not completed — Lost to Follow-up | 15 | 13 | 21

BASELINE CHARACTERISTICS:
Population: 18-45 years old Patients who underwent primary cesarean section in our hospital over 37 weeks of gestation Patients whose Pfannenstiel incision was closed subcutaneously
Groups:
- Group 1 (Vicryl Suture™(Polyglactin 910)): The group of patients who had a cesarean section for the first time and whose skin incision was closed with Vicryl suture™ (Polyglactin 910) Evaluation of wound infection at the 10th postoperative day control: Discharge, redness, increased temperature and opening were accepted as wound infection. Evaluation of the cosmetic results of the incision line in all groups at the 2nd and 6th month postoperative controls: The cosmetic results of wound healing are two different It was evaluated with a scale. The Patient and Observer Assessment Scale (POSAS) is a questionnaire developed to evaluate scar quality. The researcher scores six items: vascularization, pigmentation, thickness, surface roughness, elasticity, and surface area. The participant scores six items: pain, itching, color, thickness, relief, and flexibility. All items are scored on a 10-point multiple scale; 1 point is given when the scar characteristic resembles 'normal skin', and 10 points are given when it reflects the 'worst scar'. All items are summed to determine the total scar score; a higher score represents worse scar quality. The Vancouver scar scale (VSS) consists of four variables: vascularity, height (thickness), elasticity and pigmentation. The total score ranges from 0 to 14, with a score of 0 reflecting normal skin.
- Group 2 (Prolene Suture™(Polypropylene)): The group of patients who had a cesarean section for the first time and whose skin incision was closed with Prolene suture™ (polypropylene) Evaluation of wound infection at the 10th postoperative day control: Discharge, redness, increased temperature and opening were accepted as wound infection. Evaluation of the cosmetic results of the incision line in all groups at the 2nd and 6th month postoperative controls: The cosmetic results of wound healing are two different It was evaluated with a scale. The Patient and Observer Assessment Scale (POSAS) is a questionnaire developed to evaluate scar quality. The researcher scores six items: vascularization, pigmentation, thickness, surface roughness, elasticity, and surface area. The participant scores six items: pain, itching, color, thickness, relief, and flexibility. All items are scored on a 10-point multiple scale; 1 point is given when the scar characteristic resembles 'normal skin', and 10 points are given when it reflects the 'worst scar'. All items are summed to determine the total scar score; a higher score represents worse scar quality. The Vancouver scar scale (VSS) consists of four variables: vascularity, height (thickness), elasticity and pigmentation. The total score ranges from 0 to 14, with a score of 0 reflecting normal skin.
- Group 3 (Monocryl Suture™ (Polyglecaprone 25)): The group of patients who had a cesarean section for the first time and whose skin incision was closed with Tekmon suture™ (Polyglecaprone 25) Evaluation of wound infection at the 10th postoperative day control: Discharge, redness, increased temperature and opening were accepted as wound infection. Evaluation of the cosmetic results of the incision line in all groups at the 2nd and 6th month postoperative controls: The cosmetic results of wound healing are two different It was evaluated with a scale. The Patient and Observer Assessment Scale (POSAS) is a questionnaire developed to evaluate scar quality. The researcher scores six items: vascularization, pigmentation, thickness, surface roughness, elasticity, and surface area. The participant scores six items: pain, itching, color, thickness, relief, and flexibility. All items are scored on a 10-point multiple scale; 1 point is given when the scar characteristic resembles 'normal skin', and 10 points are given when it reflects the 'worst scar'. All items are summed to determine the total scar score; a higher score represents worse scar quality. The Vancouver scar scale (VSS) consists of four variables: vascularity, height (thickness), elasticity and pigmentation. The total score ranges from 0 to 14, with a score of 0 reflecting normal skin.
- Total: Total of all reporting groups
Arm/Group | Group 1 (Vicryl Suture™(Polyglactin 910)) | Group 2 (Prolene Suture™(Polypropylene)) | Group 3 (Monocryl Suture™ (Polyglecaprone 25)) | Total
Number analyzed (Participants) | 100 | 100 | 100 | 300
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.5 (5.8) | 27.3 (5.6) | 27.9 (5.7) | 27.9 (6.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 100 | 100 | 100 | 300
  Male | 0 | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
BMI [Mean (Standard Deviation); unit: kg/m²] | 29.2 (5.5) | 30.8 (5.1) | 30.4 (4.8) | 30.1 (5.8)

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of the Difference Between the Groups in the Number of Patients With Wound Infection at the End of the 10th Postoperative Day
Description: At the 10th postoperative day follow-up, discharge, redness, increased temperature and wound opening were considered as wound infection.
Time Frame: 0-10. day
Population: Inclusion Criteria:
  18-45 years old Patients who had a primary cesarean section at 37w Patients with a Pfannenstiel incision closed subcutaneously
Measure: Count of Participants; unit: Participants
Groups:
- Group 1 (Vicryl Suture™(Polyglactin 910)): The group of patients who had a cesarean section for the first time and whose skin incision was closed with Vicryl suture™ (Polyglactin 910) Evaluation of wound infection at the 10th postoperative day control: Discharge, redness, increased temperature and opening were accepted as wound infection.
- Group 2 (Prolene Suture™(Polypropylene)): The group of patients who had a cesarean section for the first time and whose skin incision was closed with Prolene suture™ (polypropylene) Evaluation of wound infection at the 10th postoperative day control: Discharge, redness, increased temperature and opening were accepted as wound infection.
- Group 3 (Monocryl Suture™ (Polyglecaprone 25)): The group of patients who had a cesarean section for the first time and whose skin incision was closed with Tekmon suture™ (Polyglecaprone 25) Evaluation of wound infection at the 10th postoperative day control: Discharge, redness, increased temperature and opening were accepted as wound infection.
Arm/Group | Group 1 (Vicryl Suture™(Polyglactin 910)) | Group 2 (Prolene Suture™(Polypropylene)) | Group 3 (Monocryl Suture™ (Polyglecaprone 25))
Number analyzed (Participants) | 92 | 95 | 96
Participants
  No wound infection | 80 | 90 | 93
  Wound infection | 12 | 5 | 3

2. Primary Outcome: Comparison of Incision Cosmetic Results Between Group 1 (Vicryl Suture™(Polyglactin 910)) and Group 2 (Prolene Suture™(Polypropylene)) at the End of the 2nd Postoperative Month and at the End of the 6th Postoperative Month by POSAS
Description: The cosmetic outcome of wound healing was assessed using two different scales. The Patient and Observer Assessment Scale (POSAS) is a questionnaire developed to assess wound quality. The investigator scores six items: vascularization, pigmentation, thickness, surface roughness, elasticity, and surface area. The participant scores six items: pain, itching, color, thickness, elevation, and elasticity. All items are scored on a 10-point scale; 1 point is given when the wound characteristic is similar to 'normal skin', and 10 points are given when it reflects the 'worst wound'. The total score closest to normal skin is 11, and the total score reflecting the worst wound is 110. The other scale is the Vancouver Wound Scale (VSS), consisting of four variables: vascularity, height (thickness), elasticity, and pigmentation. The total score ranges from 0 to 13, with 0 reflecting normal skin and 13 reflecting the worst wound.
Time Frame: End of the 2nd month and 6th month
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Group 1 (Vicryl Suture™(Polyglactin 910)): The group of patients who had a cesarean section for the first time and whose skin incision was closed with Vicryl suture™ (Polyglactin 910) Evaluation of cosmetic outcomes of the incision line in all groups at 2 and 6 months postoperatively: Cosmetic outcomes of wound healing were assessed using two different scales. The Patient and Observer Assessment Scale (POSAS) is a questionnaire developed to assess scar quality. The examiner scores six items: vascularization, pigmentation, thickness, surface roughness, elasticity, and surface area. The participant scores six items: pain, itch, color, thickness, relief, and flexibility. A score of 1 is given for all items indicating a scar characteristic similar to normal skin, and 10 for a scar characteristic reflecting the worst scar. All items are summed to determine a total scar score; a higher score represents worse scar quality. The Vancouver Scar Scale (VSS) consists of four variables: vascularization, height (thickness), elasticity, and pigmentation. The total score ranges from 0 to 14, with a score of 0 reflecting normal skin and a higher score representing worse scar quality.
- Group 2 (Prolene Suture™(Polypropylene)): The group of patients who had a cesarean section for the first time and whose skin incision was closed with Prolene suture™ (polypropylene) Evaluation of cosmetic outcomes of the incision line in all groups at 2 and 6 months postoperatively: Cosmetic outcomes of wound healing were assessed using two different scales. The Patient and Observer Assessment Scale (POSAS) is a questionnaire developed to assess scar quality. The examiner scores six items: vascularization, pigmentation, thickness, surface roughness, elasticity, and surface area. The participant scores six items: pain, itch, color, thickness, relief, and flexibility. A score of 1 is given for all items indicating a scar characteristic similar to normal skin, and 10 for a scar characteristic reflecting the worst scar. All items are summed to determine a total scar score; a higher score represents worse scar quality. The Vancouver Scar Scale (VSS) consists of four variables: vascularization, height (thickness), elasticity, and pigmentation. The total score ranges from 0 to 14, with a score of 0 reflecting normal skin and a higher score representing worse scar quality.
Arm/Group | Group 1 (Vicryl Suture™(Polyglactin 910)) | Group 2 (Prolene Suture™(Polypropylene))
Number analyzed (Participants) | 85 | 87
units on a scale
  POSAS 2nd month evaluation | 26.9 (8.9) | 20.5 (5.1)
  POSAS 6th month evaluatıon | 20.9 (6.1) | 16.5 (3.9)

3. Primary Outcome: Comparison of Incision Cosmetic Results Between Group 1 (Vicryl Suture™(Polyglactin 910)) and Group 3 (Tekmon Suture™(Poliglekapron 25)) at the End of the 2nd Postoperative Month and at the End of the 6th Postoperative Month by POSAS
Description: as for outcome 2
Time Frame: End of the 2nd month and 6thmonth
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Group 3 (Monocryl Suture™ (Polyglecaprone 25)): The group of patients who had a cesarean section for the first time and whose skin incision was closed with Tekmon suture™ (Polyglecaprone 25) Evaluation of cosmetic outcomes of the incision line in all groups at 2 and 6 months postoperatively: Cosmetic outcomes of wound healing were assessed using two different scales. The Patient and Observer Assessment Scale (POSAS) is a questionnaire developed to assess scar quality. The examiner scores six items: vascularization, pigmentation, thickness, surface roughness, elasticity, and surface area. The participant scores six items: pain, itch, color, thickness, relief, and flexibility. A score of 1 is given for all items indicating a scar characteristic similar to normal skin, and 10 for a scar characteristic reflecting the worst scar. All items are summed to determine a total scar score; a higher score represents worse scar quality. The Vancouver Scar Scale (VSS) consists of four variables: vascularization, height (thickness), elasticity, and pigmentation. The total score ranges from 0 to 14, with a score of 0 reflecting normal skin and a higher score representing worse scar quality.
Arm/Group | Group 1 (Vicryl Suture™(Polyglactin 910)) | Group 3 (Monocryl Suture™ (Polyglecaprone 25))
Number analyzed (Participants) | 85 | 79
units on a scale
  POSAS 2nd month evaluatıon | 26.9 (8.9) | 18.7 (3.9)
  POSAS 6th month evaluatıon | 20.9 (6.1) | 14.5 (2.4)

4. Primary Outcome: Comparison of Incision Cosmetic Results Between Group 2 (Prolene Suture™(Polypropylene)) and Group 3 (Tekmon Suture™(Poliglekapron 25)) at the End of the 2nd Postoperative Month and at the End of the 6th Postoperative Month by POSAS
Description: as for outcome 2
Time Frame: End of the 2nd month and 6thmonth
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Group 2 (Prolene Suture™(Polypropylene)) | Group 3 (Monocryl Suture™ (Polyglecaprone 25))
Number analyzed (Participants) | 86 | 79
units on a scale
  POSAS 2nd month evaluatıon | 20.5 (5.1) | 18.7 (3.9)
  POSAS 6sh month evaluatıon | 16.5 (3.9) | 14.5 (2.4)

5. Primary Outcome: Comparison of Incision Cosmetic Results Between Group 1(Vicryl Suture™(Polyglactin 910)) and Group 2(Prolene Suture™(Polypropylene)) at the End of the 2nd Postoperative Month and at the End of the 6th Postoperative Month by The Vancouver Scar Scale (VSS)
Description: as for outcome 2
Time Frame: End of the 2nd month and 6th month
Population: as for outcome 1
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Group 1 (Vicryl Suture™(Polyglactin 910)) | Group 2 (Prolene Suture™(Polypropylene))
Number analyzed (Participants) | 85 | 87
units on a scale
  VSS 2nd month evaluatıon | 4 [1 to 8] | 3 [1 to 5]
  VSS 6th month evaluatıon | 3 [1 to 6] | 3 [1 to 6]

6. Primary Outcome: Comparison of Incision Cosmetic Results Between Group 1(Vicryl Suture™(Polyglactin 910)) and Group 3(Tekmon Suture™(Poliglekapron 25)) at the End of the 2nd Postoperative Month and at the End of the 6th Postoperative Month by The Vancouver Scar Scale(VSS)
Description: as for outcome 2
Time Frame: End of the 2nd month and 6th month
Population: as for outcome 1
Measure: Median (Full Range); unit: units on a scale
Groups:
- Group 3 (Tekmon Suture™ (Polyglecaprone 25)): The group of patients who had a cesarean section for the first time and whose skin incision was closed with Tekmon suture™ (Polyglecaprone 25) Evaluation of cosmetic outcomes of the incision line in all groups at 2 and 6 months postoperatively: Cosmetic outcomes of wound healing were assessed using two different scales. The Patient and Observer Assessment Scale (POSAS) is a questionnaire developed to assess scar quality. The examiner scores six items: vascularization, pigmentation, thickness, surface roughness, elasticity, and surface area. The participant scores six items: pain, itch, color, thickness, relief, and flexibility. A score of 1 is given for all items indicating a scar characteristic similar to normal skin, and 10 for a scar characteristic reflecting the worst scar. All items are summed to determine a total scar score; a higher score represents worse scar quality. The Vancouver Scar Scale (VSS) consists of four variables: vascularization, height (thickness), elasticity, and pigmentation. The total score ranges from 0 to 14, with a score of 0 reflecting normal skin and a higher score representing worse scar quality.
Arm/Group | Group 1 (Vicryl Suture™(Polyglactin 910)) | Group 3 (Tekmon Suture™ (Polyglecaprone 25))
Number analyzed (Participants) | 85 | 79
units on a scale
  VSS 2nd month evaluatıon | 4 [1 to 8] | 3 [1 to 6]
  VSS 6th month evaluatıon | 3 [1 to 6] | 2 [1 to 4]

7. Primary Outcome: Comparison of Incision Cosmetic Results Between Group 2(Prolene Suture™(Polypropylene)) and Group 3(Tekmon Suture™(Poliglekapron 25)) at the End of the 2nd Postoperative Month and at the End of the 6th Postoperative Month by The Vancouver Scar Scale(VSS)
Description: as for outcome 2
Time Frame: End of the 2nd month and 6th month
Population: as for outcome 1
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Group 2 (Prolene Suture™(Polypropylene)) | Group 3 (Monocryl Suture™ (Polyglecaprone 25))
Number analyzed (Participants) | 86 | 79
units on a scale
  VSS 2nd month evaluatıon | 3 [1 to 5] | 3 [1 to 6]
  VSS 6th month evaluatıon | 3 [1 to 6] | 2 [1 to 4]

ADVERSE EVENTS:
Time Frame: 6 months
Description: Other (Not Including Serious) Adverse Events
Arm/Group | Group 1 (Vicryl Suture™(Polyglactin 910)) | Group 2 (Prolene Suture™(Polypropylene)) | Group 3 (Monocryl Suture™ (Polyglecaprone 25))
All-Cause Mortality (participants affected / at risk) | 0/85 | 0/87 | 0/79
Serious Adverse Events (participants affected / at risk) | 0/85 | 0/87 | 0/79
Other Adverse Events (participants affected / at risk) | 12/85 | 5/87 | 2/79
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Group 1 (Vicryl Suture™(Polyglactin 910)) (N=85) | Group 2 (Prolene Suture™(Polypropylene)) (N=87) | Group 3 (Monocryl Suture™ (Polyglecaprone 25)) (N=79)
dehiscence and discharge (Skin and subcutaneous tissue disorders) | 11 | 4 | 2
Apse (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hematom (Skin and subcutaneous tissue disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-02-22): https://cdn.clinicaltrials.gov/large-docs/13/NCT06119113/Prot_SAP_ICF_000.pdf